CLINICAL TRIAL: NCT06928480
Title: Effectiveness and Acceptability of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in People With Long COVID-19.
Acronym: UP-LONGCOVID-R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Hospital Royo Villanova de Zaragoza (Unknown)
Responsible Party: Principal Investigator, Jorge Javier Osma López, Principal Investigator, Associate Professor of Psychology, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UP-LONGCOVID-RCT; PROY_S22_24 (Other Grant/Funding Number: Gobierno de Aragón)
Record Dates: First submitted 2025-03-28; First posted 2025-04-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Long Covid-19; Emotional Disorder; Anxiety; Depression Disorders; Emotion Regulation
Keywords: Long COVID-19; Emotional Disorders; Emotion regulation skills; Unified Protocol; Transdiagnostic; Psychological; Cognitive Behavioral
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Anxiety Disorders; Emotional Regulation | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified Protocol Psychological Intervention (Experimental): The 45 participants assigned to this condition will receive the Unified Protocol psychological intervention through 12 sessions. Weekly session will be conducted online (via Google Meet). Each sessions will last 2 hours.
  Interventions: Behavioral: Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders
- Control Group-Waiting list (Other): The 45 participants assigned to this condition will remain as a control group on a waiting list for the 12 weeks of the program that participants in the experimental group receive.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders — This transdiagnostic psychological intervention is focused on training emotion regulation skills. This program is composed by 8 modules (core modules are 3 to 7).
  In this study we will use a group online format (videocalls). Each sessin will last 2 hours. The contents of the UP will be distributed in 12 online sessions as follows:
  * Module 1 (session 1): Setting goals and maintaining motivation.
  * Module 2 (sessions 2 and 3): Understanding your emotions.
  * Module 3 (sessions 4 and 5): Mindful Emotions Awareness.
  * Module 4 (sessions 6 and 7): Flexible thinking.
  * Module 5 (session 8): Emotional baheviors.
  * Module 6 (session 9): Facing physical sensations.
  * Module 7 (sessions 10 and 11): Emotionl exposures.
  * Module 8 (Session 12): Relapse prevention.
  Arms: Unified Protocol Psychological Intervention
Other: Treatment as Usual (TAU) — This intervention will act as a control condition. During the waiting period (12 weeks) participants assigned to this condition will continue receiving Treatment As Usual at the Royo Villanova Hospital. It consists of regular contact with doctors to monitor the physical symptomsof long COVID-19.
  After the 12 weeks, participants in this conditions will join the experimental group and they will receive the psychological intervention following the same procedure described for the experimental condition.
  Arms: Control Group-Waiting list

SUMMARY:
This Randomized Controlled Trial (RCT) aims to assess the effectiveness and acceptability of the Unified Protocol (UP) in an online group format for the treatment of emotional disorders in adults. Participants will be 90 adults (45 in the control group and 45 in the experimental group) with diagnosis of long COVID and comorbid emotional disorders. Participants will be recruited at Hospital Royo Villanova from Zaragoza, Spain.

In this study it will be explored whether the changes obtained after the intervention in emotional disorders and cognitive complaints are maintained over 12 months. Additionally, levels of chronic stress will be longitudinally evaluated in the experimental group through accumulated cortisol levels in hair, before and after the application of the UP.

DETAILED DESCRIPTION:
The COVID-19 disease has caused one of the largest pandemics in history, with significant health, social, and economic negative consequences. A significant proportion of the population has not overcome these negative consequences. It has been found that 10-20% of patients with COVID-19 do not recover their previous health status and develop persistent symptoms over time. This condition has been defined by the WHO as post-COVID-19 condition or long COVID-19, characterized by the presence of physical, cognitive, and emotional symptoms that can last for months or even years after the acute COVID-19 infection. Some of the most prevalent symptoms are fatigue, difficulty breathing, and cognitive dysfunction, in addition to significant psychological impairments. Among these, emotional disorders (ED) are the most commonly reported in this population, including anxiety disorders, depressive disorders, and related conditions.

The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP) is a transdiagnostic Cognitive Behavioral Therapy-based pychological intervention, which has proven to be effective for the treatment of emotional disorders in different populations. The UP is focused on improving emotion regulation skills.

The main objective of this randomized controlled trial is to evaluate the effectiveness and acceptability of the Unified Protocol (UP) in an online group format for the treatment of emotional disorders in 90 adults (45 in the control group and 45 in the experimental group) with long COVID and a comorbid emotional disorder. The researchers hypothesize that the application of the UP will result in a significant reduction in emotional symptoms in the experimental group, compared to the control group. To analyze this results, the evolution of symptoms (i.e., anxiety and depressive symptoms, etc.) will be assessed over time (before and after the intervention, as well as up to 12 months follow-up). Additionally, the acceptability and satisfaction of participants after receiving the UP will be analyzed, and it will be examined whether changes in emotional symptoms are associated with changes in long COVID physical symptoms. Changes in cortisol and cortisona levels will be longitudinally examined in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Residing in Autonomous Community of Aragon (Spain).
* Being at least 18 years old.
* Understanding of Spanish.
* Being diagnosed with long COVID-19: documented SARS-CoV-2 infection and persistence of symptoms beyond 12 weeks after the acute infection.
* Symptoms of depression (ODSIS≥7) and/or anxiety (OASIS≥8).
* Meeting the criteria for an emotional disorder diagnosis.
* Having access to Internet.
* Signing the informed consent.

Exclusion Criteria:

* Pre-existing emotional symptoms prior to the acute SARS-CoV-2 infection.
* Actually receiving psychological treatment.
* Having a diagnosis of severe mental disorder (e.g., personality disorder, bipolar disorder, etc.).
* Active suicidal ideation at the time of the assessment.
* Individuals on psychotropic medication must maintain their dosage throughout the study, unless medically contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
General Depression Severity and Interference Scale (ODSIS; Bentley et al., 2014. Validated in Spanish by Osma et al., 2019) | Before the treatment, after the treatment, at three points follow up (3, 6 and 12 months after the intervention ended)
  It assesses the frequency, intensity, severity and interference of depressive symptomatology through 5 items. total scores range from 0 to 20 points, higher scores indicating more severe depressive symptoms.
General Severity and Interference Scale for Anxiety (OASIS; Norman et al., 2006. Validated in Spanish by Osma et al., 2019) | Before the treatment, after the treatment, at three points follow up (3, 6 and 12 months after the intervention ended)
  It consiste of 5 items that assess the frequency, intensity, severity and interference of anxious symptomatology. Total scores range from 0 to 20 points, higher scores represent more severe anxiety symptoms.

SECONDARY OUTCOMES:
Memory Failures of Everyday, MFE (Sunderland et al., 1983; Montejo et al., 2014) | Before the treatment, after the treatment, at three points follow up (3, 6 and 12 months after the intervention ended)
  It assesses the frequency of forgetfulness and memory lapses in daily life. Errors include forgetting names, misplacing objects, difficulties in planning, or lapses in attention.
Multidimensional Inventory for Emotional Disorders (MEDI; Rosellini and Brown, 2019. Validated in Spanish by Osma et al., 2023) | Before the treatment, after the treatment, at three points follow up (3, 6 and 12 months after the intervention ended)
  It is composed by 49 items that evaluates the transdiagnostic profile of Emotional Disorders, which is composed of nine dimensions: neurotic temperament, positive temperament, depressed mood, somatic anxiety, arousal activation, social anxiety, intrusive cognitions, traumatic re-experiencing, and avoidance.
Emotional Regulation Difficulties Scale (DERS; Gratz and Roemer, 2004. Validated in Spanish by Hervás & Jódar, 2008) | Before the treatment, after the treatment, at three points follow up (3, 6 and 12 months after the intervention ended)
  Evaluation through 36 items of difficulties in emotional regulation by means of 5 subscales: lack of control, rejection, interference, inattention and emotional confusion. Higher scores indicate greater difficulties in emotion regulation.
EuroQol (Brooks, 1996. Validated in Spanish by Badia et al., 1999) | Before the treatment, after the treatment, at three points follow up (3, 6 and 12 months after the intervention ended)
  It is composd by 5 items assessing self-perceived health status. Higher scores indicate better quality of life.
Distress Tolerance Scale (DTS; Sandín et al., 2017) | Before the treatment, after the treatment, at three points follow up (3, 6 and 12 months after the intervention ended)
  This scale evaluates, through 15 items, distress tolerance in the following dimensions: 1) Tolerance: perceived ability to tolerate emotional distress; 2) Appraisal: subjective assessment of distress; 3) Absortion: attention absorbed by negative emotions; 4) Regulation: strategies to alleviate distress.
Perceived Stress Scale (PSS; Remor y Carrobles, 2001) | Before the treatment, after the treatment, at three points follow up (3, 6 and 12 months after the intervention ended)
  This scale consists of 14 items designed to measure the level of perceived stress in daily life over the past month. The items are rated from 0 to 4, where 0 is "never" and 4 is "very often." Higher total scores indicate greater perceived stress.
An adaptation of Client Satisfaction Questionnaire (CSQ-8) of Larsen et al., 1979) | After the treatment is applied (post-assessment; approximately 12 weeks after the intervention starts)
  the adaptation made for this study includes 6 of the 8 items of the CSQ-8 (perceived quality, adequacy to previous expectations, recommendation of the treatment to friends or family, usefulness of the techniques learned, general satisfaction with the intervention and probability that they will choose an intervention of this type again) and one additional item related to the discomfort generated by the intervention. Likewise, a change has been made in the Likert response scale from 4 points in the original (0 = "Bad / Not at all" to 4 = "Excellent/Very Much") to 11 in the current one (0 = "Bad / Not at all to 10 = "Excellent/Very Much"). Higher scores represent greater satisfaction with the treatment.
Evaluation questionnaire of the UP modules (Ad hoc) | After the treatment is applied (post-assessment; approximately 12 weeks after the intervention starts)
  This questionnaire has been elaborated ad hoc. It is composed of 7 questions; one general question that evaluates the usefulness of the program to improve emotional regulation and six specific questions that separately evaluate the usefulness of each of the techniques that are worked on in the different modules of the UP to better regulate emotions . The response scale ranges from 0 (not at all) to 10 (very much). Higher scores represent higher satisfaction with the treatment.
Montreal Cognitive Assessment (MoCA; Nasreddine et al., 2005) | Only in the experimental group: Before the treatment; at two points follow up (3 and 12 months after the intervention ended)
  Brief neuropsychological test designed to assess mild cognitive impairment. It evaluates multiple cognitive domains, including visuospatial skills, memory, working memory, attention, concentration, language, executive functions, and orientation. It has a maximum score of 30 points, with a common cutoff score of 25 to identify potential cognitive deficits. A score of 25 or lower is considered indicative of cognitive impairment.
Digit Symbol subtest-Wechsler Adult Intelligence Scale-III (WAIS-III; Wechsler, 1997) | Only in the experimental group: Before the treatment; at two points follow up (3 and 12 months after the intervention ended)
  This cognitive test presents a coding matrix in which the digits from 1 to 9 are paired with a symbol. On the same sheet, a series of digits is displayed with a blank space where participants must draw the corresponding symbol. The task must be completed as quickly as possible, with a 120-second limit to match the symbols with their respective numbers. If participants fail to complete the first four lines within the allotted time, they are given additional time to ensure they gain enough experience with the digit-symbol association. The tota score is based on the number of symbols correctly paired within 120 seconds (maximum score: 133). Immediately after completing the task, the researcher provides the participant with a new sheet containing the digits from 1 to 9 arranged in two lines. In this second part, participants must complete the blank spaces by drawing from memory the symbols corresponding to each number, with no time limit.
Digit subtest from Wechsler Adult Intelligence Scale-IV (WAIS-IV; Wechsler, 2008) | Only in the experimental group: Before the treatment; at two points follow up (3 and 12 months after the intervention ended)
  The direct order digit task of this subtest evaluates verbal short-term memory and consists of a numeric recall task that measures the mechanical repetition of a sequence of numbers. The reverse order digit task assesses verbal working memory and requires participants to recall a sequence of numbers in reverse order (maximum score: 9). The memory capacity evaluated with these two tasks is defined as the longest sequence that participants can repeat without errors, allowing two attempts for each sequence length (maximum score: 8).
Cortisol and cortisona levels | Only in the experimental group: Before the treatment; at two points follow up (3 and 12 months after the intervention ended)
  Hair sample will be collected from the posterior vertex or nape area, where growth is continuous and less exposed to contaminants. For this, a small portion of hair will be tied with thread near the cut area, which will allow identification of the portion closest to the scalp at the time of analysis and prevent hair loss. Using clean scissors, the hair will be cut as close as possible to the scalp, obtaining a segment of approximately 3 cm in length. This will allow for the evaluation of cortisol levels accumulated over the last three months, as hair grows on average 1 cm per month.

OTHER OUTCOMES:
Structured interview for anxiety disorders and related disorders, according to the DSM-5 (ADIS-5; Brown & Barlow, 2014) | Before the treatment is administered to determine inclusion criteria (approximately 2 weeks before the interventions starts)
  Diagnostic interview to determine the clinical diagnosis of emotional disorder (ED). The following diagnoses according to the DSM-V are included within the category of emotional disorder: major depressive disorder, dysthymic disorder, panic disorder, agoraphobia, obsessive-compulsive disorder, generalized anxiety disorder, post-traumatic stress disorder, social anxiety disorder, hypochondria, and adjustment disorders. Patients with anxiety disorders not otherwise specified and those with depressive disorders not otherwise specified will also be included in the study.
Sociodemographic information | Before the treatment is administered to characterize the sample (approximately 2 weeks before the interventions starts).
  Ad hoc questionnaire to assess:
  Sex, age, place of residence, marital status, employment status, lifestyle habits (smoking, alcohol, physical activity, diet), vaccination against SARS-CoV-2 information.
Long COVID-19 pre-assessment questionnaire | Before the treatment is administered to characterize the sample (approximately 2 weeks before the interventions starts).
  This questionnaire is designed to assess the symptoms and impact of long COVID-19 symptoms on patients' daily lives. It evaluates information about physical and cognitive function as well as levels of fatigue and COVID-19 infection history.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Royo Villanova, Zaragoza, Zaragoza
  - Hospital Royo Villanova, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Access Criteria: Under reasonable request.